CLINICAL TRIAL: NCT05102058
Title: Magnesium and Dexmedetomidine Combination Reduces Sodium Nitroprusside Requirement in Laparoscopic Pheochromocytoma
Brief Title: Magnesium and Dexmedetomidine in Pheochromocytoma
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nukhet Sivrikoz, Attending Anesthesiologist, Istanbul University
Other Study IDs: 2021/42
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Phaeochromocytoma Crisis; Hemodynamic Instability
Keywords: Magnesium; Dexmedetomidine; Nitroprusside; Pheochromocytoma
MeSH Terms: conditions — Pheochromocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional group (GC): Not receive perioperative additional medication.
- Magnesium-dexmedetomidine therapy group (GMD): Received oral 300 mg magnesium one week before surgery and magnesium-dexmedetomidine combination perioperatively.
  Interventions: Drug: Magnesium-Dexmedetomidine

INTERVENTIONS:
Drug: Magnesium-Dexmedetomidine — Received oral 300 mg magnesium one week before surgery and magnesium-dexmedetomidine combination perioperatively
  Groups: Magnesium-dexmedetomidine therapy group (GMD)

SUMMARY:
Anesthesia management of pheochromocytoma excision surgery is associated with severe hemodynamic fluctuations.The objective of this study was to compare the hypertensive episodes requiring sodium nitroprusside administration between the group treated with magnesium-dexmedetomidine and conventional group in pheochromocytoma.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification (ASA) 1-3
* high urinary catecholamine or metabolites
* tumor sizes < 5 cm
* body mass index (BMI) <35 kg/m2

Exclusion Criteria:

* open surgery
* bilateral masses
* tumor larger than 5 cm
* incomplete data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' data who were aged 18-75, had the American Society of Anesthesiologists classification (ASA) 1-3 and high urinary catecholamine or metabolites. Patients with tumor sizes < 5 cm and body mass index (BMI) <35 kg.m-2 were examined, who were evaluated according to Endocrine Society Practice Guideline and provided the Roizen criteria.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Sodium nitroprusside (SNP) requirement | intraoperative period
  intraoperative hypertensive episodes requiring SNP therapy

SECONDARY OUTCOMES:
vasoactive therapy | intraoperative period
  hemodynamic fluctuations (hypotension, tachycardia, severe hypertensive crisis) which needed vasoactive therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nükhet Sivrikoz, MD, Principal Investigator — Attending anesthesiologist